CLINICAL TRIAL: NCT00087789
Title: A Phase I, Dose-Escalating Study to Assess the Safety and Tolerability of CERE-110 [Adeno-Associated Virus (AAV)-Based Vector-Mediated Delivery of Beta-Nerve Growth Factor (NGF)] in Subjects With Mild to Moderate Alzheimer's Disease
Brief Title: CERE-110 in Subjects With Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sangamo Therapeutics (Industry)
Collaborators: Ceregene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CERE-110-01
Record Dates: First submitted 2004-07-13; First posted 2004-07-16 (Estimated); Last update posted 2022-11-10 (Actual); Status verified 2016-10

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; Gene Transfer
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: CERE-110: Adeno-Associated Virus Delivery of NGF — CERE-110 2.0 x 10^10 vg, CERE-110 1.0 x 10^11 vg, CERE-110 2.0 x 10^11 vg

SUMMARY:
This is a Phase I clinical study to assess the safety, tolerability and biologic activity of in vivo AAV-mediated delivery of CERE-110. Up to 12 subjects will receive open label CERE-110 in dose-escalating fashion. All subjects will receive bilateral, stereotactic injections of CERE-110 for a total of four (Dose A and B) and six (Dose C) injections to target the basal forebrain region of the brain containing the nucleus basalis of Meynert (NBM). All study participants will be observed for a 24-month period and then followed annually.

ELIGIBILITY:
Inclusion Criteria:

* Alzheimer's disease as determined by NINCDS/ADRDA criteria.
* Score of ≤ 4 on a modified Hachinski Ischemia Scale
* Mini-Mental State Exam (MMSE) score in the range of 16 to 28, inclusive
* No significant neurological or medical abnormalities contraindicating surgery, MRI/PET imaging or study participation
* Subjects stable on standard-of-care medications (i.e., acetylcholinesterase inhibitors) for Alzheimer's disease for 3 months prior to entry
* A Hamilton Depression Scale score of ≤ 12 on a 17-item scale and no history of major depressive episode within the last 2 years
* A score of < 15 on the Beck Depression Inventory
* Adequate visual and auditory acuity to allow neuropsychological testing
* Good health with no clinically significant medical or psychological conditions
* An MRI of the head at screen that is negative for evidence of infection, tumor, infarction or other focal (e.g., subdural hematoma) or generalized lesions(e.g., v hydrocephalus) and without clinical symptoms suggestive of intervening neurological disease
* Normal serum B12, thyroid function tests, and negative syphilis antibody test
* The informed consent document must be signed by both:

a competent and willing subject, and a surrogate identified by the participant, or a legally authorized power of attorney for Health Care, or a family member

Exclusion Criteria:

* History of cancer within the last five years, except superficial basal or squamous cell skin cancer or cervical carcinoma in situ
* History of alcohol abuse or dependence within the last two years
* Liver serum transaminases (AST and/or ALT) > 5 times the upper limit of normal; total and/or direct bilirubin > 1.5 mg/dL, hemoglobin < 9mg/dL; PT and PTT > 2 times the upper limit of normal; creatinine clearance < 30 mL/min; positive serology for HBV or HCV; absolute neutrophil count < 1,500 cells/mm3 and a platelet count < 100,000/mm3
* Any significant systemic illness, unstable or severe medical condition(s) that could put the subject at risk during the study, interfere with outcome measures or affect compliance with the protocol procedures
* Centrally active beta-blockers, anti-Parkinsonian medications, psychostimulants, antipsychotics, neuroleptics, or narcotic analgesics, long-acting benzodiazepines or barbiturates, hypertensive agents with a CNS effect, short-acting anxiolytics or sedative hypnotics more frequently than two times per week within 14 days of screening, herbal products for Alzheimer's disease, antidepressants with significant cholinergic side effects (e.g., tricyclics), initiation or change in dose of standard treatment for Alzheimer's disease
* Other medication with significant cholinergic or anticholinergic side effects
* Warfarin (coumadin), nonsteroidal anti-inflammatory drugs, aspirin, Prozac, or Ginkgo biloba within 14 days of surgery
* Subjects who have received investigational agents or been exposed to investigational devices for 30 days prior to enrollment
* Subjects with a history of receiving gene transfer products of any kind
* Subjects who cannot undergo MRI or PET screening

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2004-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of three different doses of CERE-110 in subjects with mild to moderate Alzheimer's disease | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Joao Siffert, M.D., Study Director — Ceregene
Locations (2):
- United States (2):
  - University of California San Diego, San Diego, California
  - Rush University Medical Center, Chicago, Illinois